CLINICAL TRIAL: NCT02626988
Title: The Role of Agricultural Biodiversity in The Diet: a Vietnamese Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioversity International (Other)
Collaborators: University Ghent (Other); HealthBridge (Unknown); Center for Agriculture and Ecological Studies (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BIOHTDIET2015JR
Record Dates: First submitted 2015-12-03; First posted 2015-12-10 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Food Intake; Biodiversity
Keywords: Diet Diversity; Biodiversity; Agrobiodiversity; Nutrition; Vietnam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The intervention group will receive capacity building sessions on the 'Promotion of a biodiverse diet' and will include both Agriculture and Nutrition topics, in addition to access to routine health and nutrition checks, and agriculture extension as offered by commune and provincial staff as normal. 5 Sessions will be held in each village over 12 months.
  Interventions: Behavioral: Promotion of a biodiverse diet
- Control (No Intervention): The control group will continue to receive routine health check and nutrition education from health staff at commune health facilities. Access to agriculture extension services as offered by provincial staff will also continue as normal.

INTERVENTIONS:
Behavioral: Promotion of a biodiverse diet — Nutrition education combined with Agriculture Capacity building focused on a key set of nutritious crops. Component (C) 1 - Participatory Identification of Intervention Approach (PIIA); C2 - Local stakeholder consultation; C3 - Sensitisation of community; C4 - Formation of Diversity club. Club will receive capacity building from a Village health worker. The following topics will be covered species selected for promotion: 1. Where to locally source inputs and expected price, 2. How/when to prepare plots using organic inputs, 3. Planting and best-practice management practices, 4. Seed saving and storage and 4. Active Cooking demonstrations and Nutrition Education and counselling including Diversified cooking practices
  Arms: Intervention

SUMMARY:
What is the role of Agricultural biodiversity in improving diet diversity, quality and nutrition?

DETAILED DESCRIPTION:
Agricultural biodiversity can have an important role in improving diet diversity, quality and nutrition and can be seen as the foundation of the food and nutrition value chain.

Increasing the availability and access to local agricultural and/or wild biodiversity genetic resources has the potential to increase production, making more food available for consumption as long as entitlements to access it exist. However, as the history of food security interventions has shown, increasing the production and supply of staple crops alone is not enough to improve food security or nutritional status. However, while agricultural diversification is an important component, it is not alone sufficient to improve diet diversity. Other system elements including women's education and knowledge, intra-household dynamics and women's status and cultural beliefs and practices that improves children's health and nutrition are important to ensure biodiversity has a successful role in improving dietary diversity and quality.

ELIGIBILITY:
Inclusion Criteria:

* Woman of reproductive age (between 15-49 years) who are the mother or primary caregiver of a child between 12 and 23 months of age.
* Both the woman and the child should be permanent residents in the village selected and do not temporarily migrate outside the village cluster during the year.
* Reside in a Thai Village

Exclusion Criteria:

* Reside in a village that is the Urban center of commune/province
* Currently engaged in other agriculture or nutrition programme or Intervention apart from what is offered by government extension workers

Ages: 12 Months to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Mean intakes (g) of Dark Green leafy vegetables, Vitamin A Rich Fruit and Vegetable and Legumes, nuts and seeds | 12 months
  Mean intakes (g) of Dark Green leafy vegetables, Vitamin A Rich Fruit and Vegetable and Legumes, nuts and seeds by mothers and young children. Collected through administration of 24hour dietary recall
Proportion of women and children consuming Dark Green leafy vegetables, Vitamin A Rich Fruit and Vegetable and Legumes, nuts and seeds by mothers and young children | 12 months
  Proportion of women and children consuming Dark Green leafy vegetables, Vitamin A Rich Fruit and Vegetable and Legumes, nuts and seeds by mothers and young children. Collected through administration of 24hour dietary recall
Proportion of women and children reaching EAR of iron and vitamin A | 12 months
  Proportion of women and children reaching EAR of iron and vitamin A. Collected through administration of 24hour dietary recall
Mean species richness consumed daily | 12 months
  Mean species richness consumed daily. Collected through administration of 24hour dietary recall

SECONDARY OUTCOMES:
Proportion of women and children reaching EAR of 16 key nutrients | 12 months
  Proportion of women and children reaching EAR of 16 key nutrients. Collected through administration of 24hour dietary recall
Nutritional Knowledge of Women, score | 12 months
  Nutrition Knowledge Score. Collected through a Questionnaire.
Individual Dietary Diversity Score - Women - Score constructed of number of food groups consumed out of 10 | 12 months
  Individual Dietary Diversity Score of women. Score constructed of number of food groups consumed out of 10. Collected through administration of 24hour dietary recall
Individual Dietary Diversity Score - Children. Score constructed of count of number of food groups consumed out of 7 | 12 months
  Individual Dietary Diversity Score children. Score constructed of count of number of food groups consumed out of 7.Collected through administration of 24hour dietary recall
Minimum Dietary Diversity - Women - Proportion of women that consumed 5 or more food groups (out of 10). | 12 months
  Proportion of women that consumed 5 or more food groups (out of 10). Collected through administration of 24hour dietary recall
Minimum Dietary Diversity - Children - Proportion of children that consumed 4 or more food groups (out of 7). | 12 months
  Proportion of children that consumed 4 or more food groups (out of 7). Collected through administration of 24hour dietary recall
Child nutritional status - Wasting/Overweight - Mean change from baseline in weight-for-height Z-scores. The following measurements will be directly collected Height/Length (cm) and Weight (Kg) | 12 months
  Wasting/Overweight - Mean change from baseline in weight-for-height Z-scores. The following measurements will be directly collected Height/Length (cm) and Weight (Kg) and used to calculate the final indicator
Child nutritional status - Stunting - Mean change from baseline in height-for-age Z-scores The following direct measurements will be collected Age (months), Height/Length (cm) | 12 months
  Stunting - Mean change from baseline in height-for-age Z-scores The following direct measurements will be collected Age (months), Height/Length (cm) and used to calculate the final indicator.
Child nutritional status - Underweight - Mean change from baseline in weight-for-age Z-scores The following direct measurements will be collected Age (months) and Weight (Kg) | 12 months
  Underweight - Mean change from baseline in weight-for-age Z-scores The following direct measurements will be collected Age (months) and Weight (Kg) and used to calculate the final indicator
Mean daily intakes (g) of processed foods and drinks | 12 months
  Mean daily intakes (g) of processed foods and drinks. Collected through administration of 24hour dietary recall
Mean proportion of daily energy, fat, salt and sugar intakes from processed foods | 12 months
  Mean proportion of daily energy, fat, salt and sugar intakes from processed foods. Collected through administration of 24hour dietary recall

CONTACTS AND LOCATIONS:
Overall Officials: Jessica E Raneri, Principal Investigator — Bioversity International
Locations (1):
- Jessica E Raneri, Mai Sơn, Sơn La Province, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data will be made publically available upon publication of research results. It will be made available on the BioversityDataverse website. It will be anonymized.
Supporting Information: Study Protocol, SAP
Time Frame: within 2 years of collection of endline data
Access Criteria: Agrees to open access license